CLINICAL TRIAL: NCT07065682
Title: Effetivity of Dutasteride and Aloe Vera Extract Combination on Angiogenesis and Obstruction on Benign Prostatic Hyperplasia
Acronym: ALOE-DUTA-BPH
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Universitas Diponegoro (Other)
Responsible Party: Principal Investigator, Achmad Rizky Herda Pratama, dr. Achmad Rizky Herda Pratama, Sp.U, S.H., Universitas Diponegoro
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22010119510006
Record Dates: First submitted 2025-07-03; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: BPH (Benign Prostatic Hyperplasia)
Keywords: Aloe Vera; Benign prostate hyperplasia; VEGF; Prostate; dutasteride; uroflowmetry; prostatic hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Dutasteride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dutasteride 0,5 mg/day + Aloe Vera Extract 380 mg/day (Experimental)
  Interventions: Drug: Aloevera + dutasteride
- Dutasteride (Active Comparator): Control
  Interventions: Drug: Dutasteride (0.5mg)

INTERVENTIONS:
Drug: Aloevera + dutasteride — Dutasteride 0,5 mg/day + Aloe Vera Extract 380 mg/day
  Arms: Dutasteride 0,5 mg/day + Aloe Vera Extract 380 mg/day
Drug: Dutasteride (0.5mg) — Control
  Arms: Dutasteride

SUMMARY:
This study is a double blinded RCT with pre-post test design on the effect of combination of dutasteride and aloe vera, compared to dutasteride only, on uroflowmetry results, prostate volume, and VEGF serum level among patients with benign prostate hyperplasia. The treatment was given for 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with BPH clinically or radiologically (prostate volume > 30 gram, Qmax <15 mL/s)
* Willing to participate to the study

Exclusion Criteria:

* Clinically or radiologically suspected of having prostatic cancer
* Previous prostatic surgery
* Patients with urinary retention
* Patients with BPH complications: urinary tract infections, urolithiasis, or hydroneprhosis
* Previously consumed alpha blocker or 5ARI in the last 6 months
* Have consumed aloe vera extract routinely

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Uroflowmetry result | 12 weeks
  Qmax of Uroflowmetry result

SECONDARY OUTCOMES:
Prostatic volume | 12 weeks
  Measured by transabdominal ultrasonography
VEGF | 12 weeks
  serum VEGF level

CONTACTS AND LOCATIONS:
Locations (1):
- RSUD Karawang, Karawang, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nugroho E, Azhar A, Gunadi E. Relationship between Prostate Volume and International Prostate Symptom Score (IPSS) Degree of Tamed Prostate Enlargement on Transabdominal Ultrasonography (TAUS) and Transrectal Ultrasonography (TRUS) Examination. Biomed J Indones. 2021;1(7):112-7